CLINICAL TRIAL: NCT01100021
Title: A Phase 1, Single-centre, Double-blind, Randomized, Placebo-controlled, Two-cohort, Two-period Crossover Study of the Hemodynamic Interactions Between Avanafil and Two α-Adrenergic Blockers, Doxazosin and Tamsulosin, in Middle-aged Healthy Male Subjects
Brief Title: Hemodynamic Study of Avanafil and Two α-Adrenergic Blockers,Doxazosin and Tamsulosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wes Day, PhD/VP of Clinical, Vivus, Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TA-017
Record Dates: First submitted 2010-01-20; First posted 2010-04-08 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tamsulosin; avanafil; Doxazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- tamsulosin + avanafil (Experimental)
  Interventions: Drug: Tamsulosin and avanafil
- Doxazosin + avanafil (Experimental)
  Interventions: Drug: Doxazosin and avanafil

INTERVENTIONS:
Drug: Tamsulosin and avanafil — tamsulosin - 0.4mg daily for 18 days; avanafil - 200 mg 1 x 2 days
  Arms: tamsulosin + avanafil
Drug: Doxazosin and avanafil — doxazosin - 1 mg 1 x 1 day; 2 mg 1 x 2 days; 4 mg 1 x 4 days; 8 mg 1 x 11 days; avanafil - 200 mg 1 x 1 day
  Arms: Doxazosin + avanafil

SUMMARY:
The purpose of this study is to see if avanafil causes any changes in blood pressure and pulse rate when taken with doxazosin or tamsulosin.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent.
2. Adult male subjects 40 to 65 years of age, inclusive.
3. A body weight of at least 50 kg and a body mass index (BMI) between 18 and 32 kg/m2, inclusive [BMI will be calculated as weight in kg/(height in m)2].
4. Subjects are able to communicate with the Investigator, and to understand and comply with all requirements of study participation.
5. Medically healthy, with no clinically significant screening results (e.g., laboratory profiles, medical histories, ECGs, physical exam, etc.), in the opinion of the Investigator in consultation with the Sponsor.
6. Male subjects should be willing to use a condom and spermicide during sexual activity for 90 days after last dosing of avanafil and be willing to not donate sperm for 90 days after dosing.

Exclusion Criteria:

1. A history or presence of significant cardiovascular (including thromboembolic disorders), neurological, hematological, psychiatric, hepatic, gastrointestinal, pulmonary, endocrine, immunologic or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs or place the subjects at increased risk as determined by the Investigator.
2. Any clinically significant laboratory abnormalities as judged by the Investigator. Inclusion of a subject with out of normal range laboratory values must be approved by VIVUS prior to subject enrollment.
3. A predisposition to priapism, such as subjects with sickle cell disease or blood dyscrasias.
4. Known history of cardiovascular or cerebrovascular event, any history of angina.
5. Subjects with episode(s) of fainting or vasovagal hypotension.
6. History or ECG evidence of any high-risk arrhythmia or ECG judged by the Investigator to be clinically significant.
7. Hypertrophic obstructive or other clinically significant cardiomyopathy, moderate or severe cardiac valvular disease.
8. Subjects whose pulse is lower than 55 bpm at screening or 50 bpm prior to dosing.
9. Acute illness, especially any infection, within 2 weeks of dosing.
10. Systolic blood pressure < 90 or >150 mmHg; diastolic blood pressure < 50 or > 95 mmHg at screening or at check-in on Day -1 (2 rechecks are allowed).
11. Subjects with benign prostatic hyperplasia or orthostatic hypotension (as evidenced by reduction of 20 mmHg or more in systolic blood pressure, reduction of 10 mmHg or more in diastolic blood pressure, or evidence of cerebral hypoperfusion upon standing from a seated position).
12. History of retinitis pigmentosa or nonarteritic anterior ischemic optic neuropathy.
13. Any history of bipolar disorder or psychosis, history of psychiatric hospitalization, greater than one lifetime episode of major depression.
14. Hemoglobin < 12.0 g/dL.
15. Subjects with liver function tests > 1.5 ULN
16. Positive urine drug test and/or positive urine alcohol test at screening or at check-in on Day -1.
17. Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV) at screening.
18. Any history or presence of alcoholism or drug or substance abuse within 18 months or as defined by the Investigator.
19. Allergy to or previously significant adverse events with PDE5 inhibitors, doxazosin and tamsulosin or their constituents.
20. Use of any prescription or over-the-counter (OTC) medication, including herbal products, within the 14 days prior to Day 1. Up to 2 g per day of acetaminophen is allowed at the discretion of the Investigator.
21. Use of any drug in Appendix 1 (drugs known to have clinical significance in inhibiting or inducing liver enzymes involved in drug metabolism [CYP P450]) within 30 days prior to Day 1.
22. Blood donation or significant blood loss within 56 days prior to Day 1.
23. Plasma donation within 14 days prior to Day 1.
24. Any use of tobacco or nicotine products within 6 months prior to Day 1. Serum cotinine levels <10 ng/mL are considered to be consistent with no active smoking.
25. Any subject who received an investigational drug within 30 days or six half-lives, whichever is longer, prior to Day 1.
26. Evidence of any clinically significant medical, psychiatric, social or other condition by history, physical examination or laboratory studies that, in the opinion of the Investigator, would contraindicate the administration of study medications, affect compliance, interfere with study evaluations, limit study participation, or confound the interpretation of study results.
27. Involvement in the planning and conduct of the study (applies to both VIVUS or designee staff, or staff at the investigational site).
28. Previously participated in a trial with avanafil.

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The maximum decrease in blood pressure after dosing | 30, 20, 10 min predose; 15, 30, 45, 60, 75, 90, 105, 120 min, 2.5, 3, 3.5, 4, 5, 6, 7, 10, 12, 18, and 24 hrs postdose

SECONDARY OUTCOMES:
The maximum decrease in blood pressure and pulse rate after dosing | 30, 20, 10 min predose; 15, 30, 45, 60, 75, 90, 105, 120 min, 2.5, 3, 3.5, 4, 5, 6, 7, 10, 12, 18, and 24 hrs postdose

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sharples, MD, Principal Investigator — MDS Pharma Services, Inc
Locations (1):
- MDS Pharma Services Inc.,, Tempe, Arizona, United States